CLINICAL TRIAL: NCT06403540
Title: The Impact of Laparotomy and Analgesia Methods on Postoperative Diaphragm Muscle Contraction in Major Abdominal Surgeries.
Brief Title: The Impact of Laparotomy and Analgesia Methods on Diaphragm
Status: Recruiting | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Fethi Gultop, Principal Investigator, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 02fg
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Neoplasms; Gastrectomy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- diaphragm contraction fraction: Diaphragm muscle contraction fraction measured before and after surgery
  Interventions: Diagnostic Test: ultrasonography

INTERVENTIONS:
Diagnostic Test: ultrasonography — Using ultrasonography to measure diaphragm thickness

SUMMARY:
Major abdominal surgeries are traditionally performed via laparotomy. Analgesia is routinely administered during the postoperative period. The goal is to investigate the effects of laparotomy and analgesia methods on diaphragm function.

DETAILED DESCRIPTION:
Laparotomy is typically performed through a midline incision during major abdominal surgeries. Patients have difficulty breathing deeply after surgery, particularly because of pain. Intravenous drug administration, epidural catheter placement, and abdominal plane blocks are common methods of analgesia. In this study, the investigators will measure the diaphragm muscle thickness at the xiphoid level at the anterior axillary line in the supine position in participants who underwent laparotomy before and one hour after the operation, using ultrasonography M mode during inspiration, expiration, and forced inspiration. the investigators will test the effects of analgesia methods on diaphragm contraction in participants undergoing laparotomy.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years,
* major abdominal surgery cases

Exclusion Criteria:

* body mass index (BMI) >35 kg/m2
* illiteracy,
* communication issues,
* neuromuscular disorders,
* Advanced chronic respiratory disease,
* Previous abdominal or thoracic surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for major abdominal surgery due to gastrointestinal tumor
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
The impact of laparotomy on diaphragm thickness. | Measurement at the 1st postoperative hour
  Comparison of diaphragm muscle measurements before and after surgery

SECONDARY OUTCOMES:
The effect of analgesia methods on diaphragm thickness in patients undergoing laparoscopic surgery. | Measurement at the 1st postoperative hour
  Comparison of diaphragm muscle measurements before and after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Taşcıoğlu City Hospital, Istanbul, Turkey (Türkiye)